CLINICAL TRIAL: NCT04507048
Title: A Multicentric Randomized Controlled Trial Comparing the Efficacy of Passive Versus Active Educational Interventions in Increasing the Ability of Laypersons in Recognizing Skin Lesions at Risk for MELAnoma
Brief Title: Passive Versus Active Educational Interventions for Melanoma Recognition
Acronym: PAMela
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, Prof.ssa Caterina Longo, Professor, Azienda USL Reggio Emilia - IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/0075289
Record Dates: First submitted 2020-02-01; First posted 2020-08-10 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Educational Problems; Melanoma (Skin)
Keywords: educational intervention; melanoma; clinical trial
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive intervention (Active Comparator): Administration of a booklet containing the explanation of 2 clinical rules for early detection of atypical melanocytic lesions: the ABCDE and the "ugly duckling" rules.
  Interventions: Other: Passive educational intervention
- Active intervention (Experimental): A standardized oral explanation will be given to the patient by a dermatologist, together with the administration of a booklet containing written information of 2 clinical rules for detection of melanoma, as the ABCDE and the "ugly duckling" rules.
  Interventions: Other: Active educational intervention

INTERVENTIONS:
Other: Active educational intervention — an active educational intervention will be provided in the experimental arm, consisting in the administration of a booklet (passive intervention) + an oral standardized explanation of the booklet given by a trained dermatologist for each center.
  Arms: Active intervention
Other: Passive educational intervention — Administration of a booklet containing the explanation of 2 clinical rules for early detection of atypical melanocytic lesions: the ABCDE and the "ugly duckling" rules.
  Arms: Passive intervention

SUMMARY:
This study evaluates the efficacy of a passive versus an active educational intervention in increasing the ability of laypersons at low risk for melanoma development, in recognizing atypical skin melanocytic lesions. Patients will be randomized (1:1) to receive the active or the passive intervention.

DETAILED DESCRIPTION:
Almost 60-70% of primary melanomas are first detected by patients or their relatives and not by physicians. Then, it appears imperative to promote public campaigns in order to increase the awareness of laypersons on the most important rules for early identification of atypical skin lesions. The two main clinical rules are:

1. ABCD rule. According to this rule, lesions characterized by one of more of the following features: Asymmetry, irregular Borders, Color variegation and Diameter larger than 6 mm, should be considered at risk for malignancy. In order to evaluate Evolution, monitoring strategies have been implemented;
2. "ugly duckling" sign. According to this rule, a suspicious lesion tends to be different from the general nevus pattern of a given patient.

The passive intervention will consist in the administration of a booklet containing the explanation of this two previous clinical rules for early detection of atypical melanocytic lesions. In the active intervention a standardized explanation will be given to the patient by a dermatologist, together with the administration of the booklet.

Efficacy will be evaluated through the completion of a specific test before, immediately after and after one month the administration of the educational intervention.

ELIGIBILITY:
Inclusion Criteria:

* no personal or family history for melanoma;
* first visit for skin examination

Exclusion Criteria:

* patients referring to know and to be already confident in the use of at least one of the tested rules.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of lesions correctly evaluated as at risk | 30 ± 2 days
  Change at t1 and t2 from baseline (t0) in lesions at risk correctly identified, comparing passive and active educational intervention arms.

SECONDARY OUTCOMES:
Rate of lesions correctly assigned to the proper risk category | 30 ± 2 days
  Change at t1 and t2 from baseline (t0) in lesions correctly assigned to the proper risk category (low, intermediate, high), comparing passive and active educational intervention arms.

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - Valeria Ciciarelli, L’Aquila, AQ
  - Mariachiara Arisi, Brescia, BS
  - Giovanni Pellacani, Modena, MO
  - Caterina Longo, Reggio Emilia, RE
  - Ketty Peris, Rome, RM
  - Simone Ribero, Turin, TO
  - Elvira Moscarella, Naples